CLINICAL TRIAL: NCT04673994
Title: Cerebrovascular Response During Interval Exercise in Chronic Stroke
Brief Title: Blood Flow Response and Acute INterval Exercise
Acronym: BRAIN
Status: Completed | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00146161
Record Dates: First submitted 2020-12-08; First posted 2020-12-17 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Stroke; High Intensity Interval Exercise
Keywords: Cerebral Blood Velocity; Cerebral Autoregulation
MeSH Terms: conditions — Stroke | interventions — Single Person

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Chronic Stroke: Individuals 40-80 years old who have had a stroke 6 months to 5 years ago.
  Interventions: Behavioral: Single, acute bout of high intensity interval exercise
- CON: Control group (CON) comprised of age- and sex-matched healthy adults.
  Interventions: Behavioral: Single, acute bout of high intensity interval exercise
- CONyoung: Healthy, young adult control group (CONyoung) who are age 18-30 years old.
  Interventions: Behavioral: Single, acute bout of high intensity interval exercise

INTERVENTIONS:
Behavioral: Single, acute bout of high intensity interval exercise — Individuals will perform a single bout of high intensity interval exercise on a seated recumbent stepper. Participants will perform the pattern of high intensity interval exercise by switching between 1-minute high intensity stepping followed by 1-minute light, active recovery stepping for a total of 10 minutes.

SUMMARY:
The objective of this project is to study the cerebrovascular response to a single bout of high intensity interval exercise (HIIT) in 25 individuals with chronic stroke compared to 25 age- and sex- matched healthy controls (CON). We will enroll 25 young healthy adults (CONyoung) as a reference group. Our hypothesis is that the cerebrovascular response in individuals with chronic stroke will be significantly lower: 1) during a single bout of HIIT, and 2) during the recovery immediately following and 30 minutes after HIIT, compared to CON.

This study has 2 visits at the University of Kansas Medical Center Research in Exercise and Cardiovascular Health Laboratory. For the first visit, we will perform questionnaires about heart health, physical activity and overall health. Participants will then complete a submaximal exercise test on a seated stepper. Participants will also have a familiarization session to practice HIIT. The second visit will include cerebrovascular measures before, during, immediately after, and 30 minutes after performing HIIT.

ELIGIBILITY:
Chronic Stroke Inclusion Criteria:

* Age 40-80 years old
* Treated for stroke 6 months to 5 years ago
* Performs <150 minutes of moderate intensity exercise per week
* Able to answer consenting questions and follow a 2-step command

Chronic Stroke Exclusion Criteria:

* Stroke etiology due to COVID-19 pathology.
* Symptoms of COVID-19 and/or Positive COVID-19 test within the past 3 months
* Unable to stand from a sitting position without physical assistance
* Recent joint replacement/surgery/poor motor control that limits ability to perform exercise on a recumbent stepper
* Insulin injection dependent diabetes
* Dependent on supplementary oxygen
* History of other neurological disease (Multiple Sclerosis, Alzheimer's disease, Parkinson's disease)
* Unable to find TCD signal on the stroke-affected or non-affected MCA.

CON Inclusion Criteria:

* Matched age ± 5 years to participant with chronic stroke
* Matched sex to participant with chronic stroke
* Performs <150 minutes of moderate intensity exercise per week
* Able to answer consenting questions and follow a 2-step command

CON Exclusion Criteria:

* Symptoms of COVID-19 and/or Positive COVID-19 test within the past 3 months
* Unable to stand from a sitting position without physical assistance
* Recent joint replacement/surgery/poor motor control that limits ability to perform exercise on a recumbent stepper
* Insulin injection dependent diabetes
* Dependent on supplementary oxygen
* History of other neurological disease (Multiple Sclerosis, Alzheimer's disease, Parkinson's disease)
* Unable to find TCD signal on the right or left MCA.

CONyoung Inclusion Criteria:

* Age 18-30 years old
* Low cardiac risk (defined by the American College of Sports Medicine)
* Able to find TCD signal on the right or left MCA

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will recruit individuals with chronic stroke, age- and sex-matched controls (CON) and young healthy controls (CONyoung) within the community.
Sampling Method: Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
Change in Middle Cerebral Artery Blood Velocity (MCAv) | Pre-to-post intervention, ~40 minutes
  blood velocity traveling through the middle cerebral artery measured using the transcranial Doppler ultrasound.

SECONDARY OUTCOMES:
Change in Dynamic Cerebrovascular Autoregulation (dCA) | Pre-to-post intervention, ~40 minutes
  Ability of the cerebrovascular system to maintain MCAv independent of changes in peripheral blood pressure. Measured using transcranial Doppler ultrasound and mean arterial pressure measured with every heart beat.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra A Billinger, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No